CLINICAL TRIAL: NCT05725265
Title: Large-area Low-level Laser Therapy for Breast Cancer-related Lymphedema: a Randomized, Placebo-controlled Study
Brief Title: LLLT for BCRL: a Randomized, Placebo-controlled Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202210064DIPD
Record Dates: First submitted 2023-01-08; First posted 2023-02-13 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Lymphedema
Keywords: Breast Cancer Lymphedema; Lymphedema; Breast cancer; Low level laser therapy
MeSH Terms: conditions — Breast Cancer Lymphedema; Lymphedema; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Large-area low-level laser therapy (Experimental): Large-area low-level laser therapy(Venusure) was administered at proximal forearm, upper arm and axillary region of affected side. The wavelength was 980±15nm, average dose was 10-40nm/cm2 and maximal output was 1000mW. Total treatment duration was 30 min and frequency was 3 sessions/week for 4 weeks.
  Interventions: Device: Large-area low-level laser therapy(Venusure)
- Conventional low-level laser therapy (Placebo Comparator): Conventional low-level laser therapy was administrated on antecubital fossa and the axilla of affected side. The wavelength was 808nm and maximal output was 60 mW. Total treatment duration was 30 min and frequency was 3 sessions/week for 4 weeks.
  Interventions: Device: Conventional low-level laser therapy

INTERVENTIONS:
Device: Large-area low-level laser therapy(Venusure) — The wavelength was 980±15nm, average dose was 10-40nm/cm2 and maximal output was 1000mW. Total treatment duration was 30 min and frequency was 3 sessions/week for 4 weeks; for a total of 12 sessions
  Arms: Large-area low-level laser therapy
Device: Conventional low-level laser therapy — The wavelength was 808 nm and maximal output was 60 mW. Total treatment duration was 30 min and frequency was 3 sessions/week for 4 weeks; for a total of 12 sessions.
  Arms: Conventional low-level laser therapy

SUMMARY:
This study is conducted to compare between efficacy of large and small area of low-level laser therapy (LLLT) in treatment of post mastectomy lymphedema. The change of severity of BCRL will be measured by the difference of circumference and skin thickness, detected by ultrasound. The influence on clinical symptoms, such as pain, shoulder mobility and hand function, are also investigated in the study.

DETAILED DESCRIPTION:
Breast cancer-related lymphedema (BCRL) is common complication after cancer treatment. The incidence of BCRL around is 16.6% (95% CI 13·6-20·2) after the diagnosis and higher among the group receiving the sentinel biopsy or axillary lymph dissection. The lymphedema arises from the accumulation of protein-rich lymph fluid in the interstitial spaces then results in chronic inflammation with symptoms of fibrosis, pain, limited range of motion or paresthesia. The BRCL is chronic and progressive condition, and the severity also changes over time. The definition and cut points of BCRL using inter-limb volume or arm circumference varied across the studies by different measure method. Currently, the International Society of Lymphology suggests calculating arm volume from circumferences through the truncated cone formula to qualify the severity. On the other hand, previous research found the skin and subcutis were thickened in the ipsilateral arm of patients with BCRL. Thus, the measurement of skin thickness using ultrasound may also practical to detect the progression of lymphedema. Except for physical change of upper limb, the symptoms of BCRL are also concerned. One of the most common morbidity is pain, mostly presenting 1 month after surgery (56.6%). Furthermore, BCRL might decrease shoulder range of motion. Previous study demonstrated that shoulder mobility was usually restricted at 1 month postoperatively and abduction and forward flexion were limited at first. Thus, functional disability may occurred and life of quality may be influenced. To evaluate the ability to perform functional activities, the Disability of Arm, Shoulder, and Hand Questionnaire (DASH) is an useful tool to assess the patients with BCRL.

Currently, although complete decongestive therapy (CDT) has been the standard therapy, there is still various type of noninvasive treatment on BCRL, for example, low-level laser therapy (LLLT). Low-level laser therapy (LLLT), also named photobiomodulation therapy (PBMT), is a conservative therapy through utilizing wave lengths of red or near infrared light between 650 and 1000 nm to stimulate wound healing and reduce inflammation, edema, and pain. Moreover, the Food and Drug Administration (FDA) approved the use of the LLLT for treatment of postmastectomy lymphedema in November 2006. Previous studies have demonstrated the effect of LLLT on BCRL with comparison to physical therapy or placebo. However, there is still limited data about the LLLT with different light area on improvement of severity and symptoms of BCRL. Therefore, this study is conducted to compare between efficacy of large and small area of low-level laser therapy (LLLT) in treatment of post mastectomy lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects, 20 years age or older, suffered from unilateral breast cancer with ipsilateral lumpectomy or mastectomy and lymph node dissection (sentinel biopsy or axillary dissection)
* Stage I or II unilateral secondary upper extremity lymphedema(as defined by the International Society of Lymphology)
* Girth≥ 2 cm circumferential difference compared with the uninvolved upper extremity at any 4 cm segment
* Able to commit to a long-term follow-up schedule

Exclusion Criteria:

* Metastatic cancer(stage IV)
* Pregnancy
* Presence of other extremity lymphedema (primary or secondary)
* History of deep vein thrombosis
* Pacemaker
* Artificial joints, implant or tattoo(area≥4 cm2) at the involved upper extremity
* Previous treatment with low-level laser therapy (within 3 months)
* Body mass index (BMI) > 35 (morbid obesity)
* High bleeding tendency(hemophilia)
* Receiving long-term steroid treatment (oral or systemic)

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Circumference discrepancy of bilateral upper arm | Day 30 (change of circumference discrepancy of bilateral upper limbs, comparing with the data in baseline) of each section
  Record the circumference of arm and forearm of involved and uninvolved upper extremity at 4 cm segment from cubital fossa and calculate the circumference discrepancy.
Circumference discrepancy of bilateral upper arm | Day 60 (change of circumference discrepancy of bilateral upper limbs, comparing with the data in baseline) of each section
  Record the circumference of arm and forearm of involved and uninvolved upper extremity at 4 cm segment from cubital fossa and calculate the circumference discrepancy.
Circumference discrepancy of bilateral upper arm | Day 120 (change of circumference discrepancy of bilateral upper limbs, comparing with the data in baseline) of each section
  Record the circumference of arm and forearm of involved and uninvolved upper extremity at 4 cm segment from cubital fossa and calculate the circumference discrepancy.

SECONDARY OUTCOMES:
visual analogue scale (VAS) | Day 30, Day 60, Day 120 (comparing with the data in baseline) of each section
  Record visual analogue scale (VAS) to rate the severity of pain. The total score ranges from 0 to 10. Higher score indicates greater pain intensity.
Range of motion of involved shoulder | Day 30, Day 60, Day 120 (comparing with the data in baseline) of each section
  involved upper extremity.
Skin thickness | Day 30, Day 60, Day 120 (comparing with the data in baseline) of each section
  Use ultrasound to measure the skin thickness of arm and forearm of involved upper extremity.
QuickDASH | Day 30, Day 60, Day 120 (comparing with the data in baseline) of each section
  QuickDASH(Quick Disabilities of Arm, Shoulder & Hand) is a questionnaire for patients presenting with self-reported disabilities of the arm, shoulder and hand. The QuickDASH contains 11-items; the score of each item ranges from 1 to 5 and total score ranges from 0 to 100. Higher score indicates greater level of disability and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Chueh-Hung Wu, PHD, Study Chair — Department of Physical Medicine and Rehabilitation, National Taiwan University Hospital, Taipei, Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DiSipio T, Rye S, Newman B, Hayes S. Incidence of unilateral arm lymphoedema after breast cancer: a systematic review and meta-analysis. Lancet Oncol. 2013 May;14(6):500-15. doi: 10.1016/S1470-2045(13)70076-7. Epub 2013 Mar 27. PMID 23540561
- [Background] Grada AA, Phillips TJ. Lymphedema: Pathophysiology and clinical manifestations. J Am Acad Dermatol. 2017 Dec;77(6):1009-1020. doi: 10.1016/j.jaad.2017.03.022. PMID 29132848
- [Background] Eyigor S, Cinar E, Caramat I, Unlu BK. Factors influencing response to lymphedema treatment in patients with breast cancer-related lymphedema. Support Care Cancer. 2015 Sep;23(9):2705-10. doi: 10.1007/s00520-015-2633-9. Epub 2015 Feb 8. PMID 25663541
- [Background] Mellor RH, Bush NL, Stanton AW, Bamber JC, Levick JR, Mortimer PS. Dual-frequency ultrasound examination of skin and subcutis thickness in breast cancer-related lymphedema. Breast J. 2004 Nov-Dec;10(6):496-503. doi: 10.1111/j.1075-122X.2004.21458.x. PMID 15569205
- [Background] Swenson KK, Nissen MJ, Ceronsky C, Swenson L, Lee MW, Tuttle TM. Comparison of side effects between sentinel lymph node and axillary lymph node dissection for breast cancer. Ann Surg Oncol. 2002 Oct;9(8):745-53. doi: 10.1007/BF02574496. PMID 12374657
- [Background] Verbelen H, Gebruers N, Eeckhout FM, Verlinden K, Tjalma W. Shoulder and arm morbidity in sentinel node-negative breast cancer patients: a systematic review. Breast Cancer Res Treat. 2014 Feb;144(1):21-31. doi: 10.1007/s10549-014-2846-5. Epub 2014 Feb 5. PMID 24496928
- [Background] Lee D, Hwang JH, Chu I, Chang HJ, Shim YH, Kim JH. Analysis of factors related to arm weakness in patients with breast cancer-related lymphedema. Support Care Cancer. 2015 Aug;23(8):2297-304. doi: 10.1007/s00520-014-2584-6. Epub 2015 Jan 10. PMID 25576430
- [Background] Smile TD, Tendulkar R, Schwarz G, Arthur D, Grobmyer S, Valente S, Vicini F, Shah C. A Review of Treatment for Breast Cancer-Related Lymphedema: Paradigms for Clinical Practice. Am J Clin Oncol. 2018 Feb;41(2):178-190. doi: 10.1097/COC.0000000000000355. PMID 28009597
- [Background] Robijns J, Censabella S, Bulens P, Maes A, Mebis J. The use of low-level light therapy in supportive care for patients with breast cancer: review of the literature. Lasers Med Sci. 2017 Jan;32(1):229-242. doi: 10.1007/s10103-016-2056-y. Epub 2016 Aug 19. PMID 27539464
- [Background] Wang Y, Ge Y, Xing W, Liu J, Wu J, Lin H, Lu Y. The effectiveness and safety of low-level laser therapy on breast cancer-related lymphedema: An overview and update of systematic reviews. Lasers Med Sci. 2022 Apr;37(3):1389-1413. doi: 10.1007/s10103-021-03446-3. Epub 2021 Nov 15. PMID 34779937
- [Background] Levenhagen K, Davies C, Perdomo M, Ryans K, Gilchrist L. Diagnosis of Upper Quadrant Lymphedema Secondary to Cancer: Clinical Practice Guideline From the Oncology Section of the American Physical Therapy Association. Phys Ther. 2017 Jul 1;97(7):729-745. doi: 10.1093/ptj/pzx050. PMID 28838217